CLINICAL TRIAL: NCT04535245
Title: Lung Clearance Measurement to Determine Pre-clinical Airway Involvement in Scleroderma Patients Without Lung Disease as a Risk Factor for Developing ILD
Brief Title: Lung Clearance Index to Identify Scleroderma Patients at Risk for ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Richard Meehan, Professsor of Medicine, National Jewish Health
Other Study IDs: HS 3471
Record Dates: First submitted 2020-08-12; First posted 2020-09-01 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LCI testing: LCI testing will be performed on all study subjects
  Interventions: Diagnostic Test: LCI testing

INTERVENTIONS:
Diagnostic Test: LCI testing — all subjects will have LCI testing then contacted via a phone interview or EMR review yearly times 5 to determine if they have subsequently developed ILD
  Other Names: no drugs will be administered

SUMMARY:
This National Jewish Health (NJH) Investigator Initiated pilot study funded by the Shah Foundation will prospectively perform a non invasive lung function test called Lung Clearance Index (LCI) to determine if 50 scleroderma patients without evidence of lung disease who have evidence of small airway inflammation or impairment to airflow are more likely to develop ILD than those with normal vales.50 subjects will be enrolled from the Rheumatology practice at NJH and followed with phone interviews or Electronic Medical Record (EMR) record review yearly times 5 to determine if they have subsequently developed evidence of ILD or pulmonary artery hypertension.

DETAILED DESCRIPTION:
50 scleroderma patients without evidence of lung disease who have been seen by an NJH Rheumatologist will be invited to participate. They will have their medical records reviewed to determine eligibility and then perform hand held spirometry and LCI testing. This measures evidence of small airway airflow obstruction and requires normal breathing while first on room air followed by inhaling a gas mixture of 100% oxygen. The Oxygen concentration in exhaled breathing and the number of breaths needed to return to room air concentration of Oxygen will be analyzed by a computer. Medical information from the EMR will be recorded and placed in a secure database, REDCap, for statistical analysis to determine if LCI results or other clinical features are predictive of which Scleroderma patients are most likely to subsequently develop evidence of Interstitial Lung disease (ILD) based upon yearly phone call interviews and EMR record reviews within 5 years of baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of systemic sclerosis (SSC) by an NJH Rheumatologist
* age 21-75
* No evidence of Scleroderma related Lung disease (ILD)
* Able to comprehend and sign an Institutional Review Board (IRB) approved consent form.

Exclusion Criteria:

* Patients without a Rheumatologists confirming a diagnosis (DX) of SSC
* Patients with evidence of lung involvement based upon; Thoracic imaging, abnormal Pulmonary Function Tests (PFTs); Forced Vital Capacity( FVC), Forced Expiratory Volume in 1 second (FEV1) or a Diffusion Capacity for Carbon Monoxide (DLCO) < the Lower Limit of Normal (LLN) or Saturation of Oxygen in arterial blood (SaO2) < 90% .
* Cardiac echocardiogram or right heart catheter evidence of Pulmonary Arterial Hypertension (PAH).
* < 21 or > 75 years of age
* Must not be pregnant or had eye surgery within 2 weeks of LCI testing
* Must be able to comprehend and sign an IRB approved consent form and complete LCI testing

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scleroderma patients without lung disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
The Utility of Lung Clearance Index Scores at predicting Interstitial Lung disease ( ILD) development within 5 years among Scleroderma patients without ILD. | 5 years after baseline testing
  Lung clearance index values (LCI) will be measured from all Scleroderma patients at baseline (normal value is < 7 ). The LCI scores from the cohort of Scleroderma patients who subsequently develop ILD based upon physician review of the EMR or phone interviews will be compared to the LCI scores from those scleroderma patients who did not develop ILD. Statistical analysis of LCI scores between both cohorts will determine the potential clinical utility of this non-invasive measurement of lung function in identifying those scleroderma patients who are at greatest risk for the subsequent development of ILD so treatment can be initiated early in their disease before irreversible pulmonary fibrosis develops.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Meehan, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No